CLINICAL TRIAL: NCT05317039
Title: Evaluation of Piezosurgical Buccal Plate Repositioning Technique for Horizontal Alveolar Ridge Augmentation Comparing Between Two Different Grafting Materials (a Randomized Clinical Trial)
Brief Title: Piezosurgical Buccal Plate Repositioning Technique for Horizontal Alveolar Ridge Augmentation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Piezosurgery_2021
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — silica-calcium phosphate nanocomposite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Group A will be treated with the buccal plate repositioning technique and grafted with SCPC.
  Interventions: Other: silica-calcium phosphate nanocomposite SCPC
- Group B (Active Comparator): Group B will be similarly managed and grafted using DFDBA
  Interventions: Other: freezed dried bone

INTERVENTIONS:
Other: silica-calcium phosphate nanocomposite SCPC — Patients will be treated with the buccal plate repositioning technique and grafted with SCPC then the grafted defect will be covered with a platelet-rich fibrin membrane.
  Arms: Group A
Other: freezed dried bone — Patients will be treated with the buccal plate repositioning technique and grafted using DFDBA. then the grafted defect will be covered with a platelet-rich fibrin membrane.
  Arms: Group B

SUMMARY:
Achieving prosthetically driven implant placement is a highly predictable treatment modality with reliable long-term results. Different surgical procedures have been used as a solution for reconstructing of the alveolar ridge with deficient volume. In the present study we demonstrate a modified alveolar ridge split technique for horizontal alveolar ridge augmentation (buccal plate repositioning technique) using the piezotome surgery. Evaluation of the effect of silica-calcium phosphate nanocomposite (SCPC) graft material versus demineralized freeze dried bone allograft (DFBA) in horizontal alveolar ridge augmentation before implant insertion will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with horizontal atrophy of the posterior mandible with pristine residual alveolar crest width from 2 to 4 mm.
* Augmented area length in the mesial-distal direction of less than 20 mm.
* Adequate physically healthy condition.

Exclusion Criteria:

* A systemic disease that would contraindicate oral surgical treatment.
* Treated patients who had undergone therapy involving radiation
* Patients who had received bone resection as part of an oncological treatment after a bone augmentation procedure.
* Patients are subjected to intravenous and/or oral bisphosphonate therapy after the bone augmentation procedure.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
change in alveolar ridge width | at baseline and 6 months
  All patients will receive a CBCT scan; immediately after surgery and at 6 months post-operatively. The images will be analyzed using OnDemand3D software (Cybermed Inc) CBCT analyzing software and compared to the pre-operative scan for alveolar ridge width evaluation.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt